CLINICAL TRIAL: NCT05724745
Title: Evaluation of 3D Magnetic Resonance Spirometry: Comparison with Spirometry in Healthy Subjects and Patients with Respiratory Pathologies (asthma, COPD, Bilateral Lung Transplant)
Acronym: gb-Spiro3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Principal Investigator, Vincent LEBON, Principal Investigator, Commissariat A L'energie Atomique
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEA 100-061; 2021-A00672-39 (Other: ANSM)
Record Dates: First submitted 2023-01-15; First posted 2023-02-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Asthma; COPD; BOS
Keywords: Lung disease; Asthma; COPD; Spirometry; MRI; 3D MR Spirometry
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Prone Position; Supine Position; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers, Asthmatic patients and COPD patients (Other): This arm of the study is essential to establish nominal flow-volume maps of nominal flow-volume curves and to determine the dependence of normal breathing on gravity and response to a bronchodilator in order to evaluate the sensitivity and specificity of the technique for the known lung diseases asthma and COPD by comparing data from healthy the data from healthy subjects with those from sick subjects.
  Interventions: Diagnostic Test: 1. Standard spirometry; Diagnostic Test: 2. 3D dynamic lung MRI at UTE in prone and supine positions; Drug: 3. Reversibility test with salbutamol; Diagnostic Test: 4. 3D dynamic lung MRI at UTE in supine and prone position

INTERVENTIONS:
Diagnostic Test: 1. Standard spirometry — Spirometry is performed in two positions (sitting and supine) and three types of breathing (spontaneous, forced and slow).
Diagnostic Test: 2. 3D dynamic lung MRI at UTE in prone and supine positions — Dynamic lung MRI is performed for 3D MR spirometry while the subject is lying prone and supine before a reversibility test with salbutamol.
Drug: 3. Reversibility test with salbutamol — Reversibility test with salbutamol administered using a pressurized metered dose bottle and an inhalation chamber at a dosage of 100 μg, 4 times (i.e., 400 μg in total).
Diagnostic Test: 4. 3D dynamic lung MRI at UTE in supine and prone position — Dynamic lung MRI is performed for 3D MR spirometry while the subject is lying prone and supine after the bronchodilatator's administration.

SUMMARY:
Spirometry is now the gold standard technique for assessing lung function in humans. From the shape of a flow-volume curve measured while the patient, trained by the practitioner, performs forced breaths, the forced vital capacity (FVC) and the forced expiratory volume in one second (FEV1) can be deduced and the pulmonologist is able to detect and characterize respiratory diseases as well as to evaluate current treatments. This technique is non-invasive and simple. It is widely available, robust, reproducible and sensitive to intervention. However, it requires proactive cooperation from the patient and only measures global pulmonary ventilation, without locoregional information.

An innovative strategy and an original study framework have been developed in the BioMaps laboratory to establish local maps of flow-volume curves across the lung and to jointly analyze ventilatory function and mechanical behavior at any point in the lung: 3D magnetic resonance spirometry. As respiratory mechanics fundamentally supports ventilatory function, this technique should open a new avenue to non-invasively explore lung function while providing a better diagnosis of regional lung diseases.

DETAILED DESCRIPTION:
Main objectiif / Evaluate the concordance of the results provided by 3D spirometry using compared with those obtained by spirometry in four populations: healthy four populations: healthy volunteers, asthma patients, patients with chronic obstructive pulmonary, chronic obstructive pulmonary disease (COPD) and lung transplant patients. with and without bronchiolitis obliterans syndrome (BOS). obliterative bronchiolitis syndrome (BOS).

ELIGIBILITY:
Inclusion Criteria:

Generic inclusion criteria

* Ability to understand the nature and objectives of the study
* Ability to remain immobile in an MRI scanner in supine position for the entire duration of the acquisitions
* Ability to give free and informed written consent Specific inclusion criteria for healthy volunteers
* Age: 18-45 years
* No known and diagnosed pulmonary pathology such as respiratory insufficiency, COPD, asthma or cancer
* Ability to remain motionless in an MRI scanner in a prone position for a total of 50 min.
* Non-smoker and non-smoker Specific inclusion criteria for asthma patients
* Age: 18-80 years
* Asthma of varying degrees of severity, depending on inhalation required to achieve control:
* Diagnosis of asthma classified as moderate according to the Global initiative for asthma (GINA) guidelines for at least 6 months
* Diagnosis of asthma classified as severe according to the Global initiative for asthma (GINA) guidelines for at least 6 months months with initiation of biotherapy planned by their pulmonologist
* Non-smoker and non-vapourist Specific inclusion criteria for COPD patients
* Age: 40-80 years
* COPD of varying degrees of severity:
* Diagnosis of COPD classified as moderate according to the Global initiative for chronic obstructive lung disease guidelines (GOLD 2: VEMS = 50-79%)
* Diagnosis of COPD classified as severe according to the guidelines for chronic obstructive lung disease (GOLD 3: VEMS = 30-49%) Specific inclusion criteria for patients with bilateral lung transplants with BOS
* Age: 18-90 years
* Irreversible FEV1 < 80% of baseline with FEV1/FVC ratio FEV1/FVC < 0.7
* Absence of visible parenchymal opacity on CT scan (non inclusion of mixed RAS/CLAD)
* Absence of significant bronchial stenosis (having required endoscopic endoscopic treatment)
* No diaphragmatic involvement (established by sniff test under fluoroscopy fluoroscopy or diaphragmatic ultrasound) Specific inclusion criteria for patients with bilateral lung transplants without BOS
* Age: 18-90 years
* FEV1 > 90% baseline for more than 24 months after the date of date of lung transplantation
* Absence of significant bronchial stenosis (requiring endoscopic endoscopic treatment)
* Absence of diaphragmatic impairment (established by sniff test under fluoroscopy or diaphragmatic ultrasound)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between (1) spontaneous expiratory volume in 1 s (SEV1) and tidal volume (TV) and (2) FEV1 and FVC | 2 months
  SEV1 and TV are extracted from the flow-volume curve calculated by integration over the whole lung of the local flow-volume curves obtained by 3D MR spirometry and FEV1 and FVC extracted from the flow-volume curve obtained by standard spirometry
Difference of expiratory volume in 1 s (SEV1) and tidal volume (TV) between the left and right lungs | 2 months
  SEV1 and TV are extracted from the integrated flow-volume curves over the left and right lungs
Difference in expiratory volume in 1 s (SEV1) and tidal volume (TV) for the anterior-posterior, inferior-superior and medial-lateral lung regions | 2 months
  SEV1 and TV are extracted from the integrated flow-volume curves over the anterior-posterior, inferior-superior and medial-lateral lung regions

CONTACTS AND LOCATIONS:
Locations (1):
- CEA | Service Hospitalier Fréderic Joliot, Orsay, France, France

IPD SHARING:
Plan to Share IPD: No